CLINICAL TRIAL: NCT00748748
Title: Effect of Lactobacillus Probiotic on Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fargo VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephanie Borchardt, Tze Shien Lo, MD, Fargo VA Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VERA 437
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Antibiotic-associated Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Lactobacillus rhamnosus GG capsule three times per day while taking their antibiotic(s) and for 7 days following completion of the antibiotic.
  Interventions: Biological: Culturelle

INTERVENTIONS:
Biological: Culturelle — 10^10 Lactobacillus rhamnosus GG per capsule

SUMMARY:
Diarrhea is a common side effect of antibiotics; it may prolong hospital stay, increase the risk of other infections, develop into more serious forms of disease, and lead to premature discontinuation of the needed antibiotic. The purpose of this study is to examine the safety and effectiveness of a capsule containing Lactobacillus rhamnosus GG in the prevention of diarrhea associated with antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Participants (male or female inpatients) 18 to 64 years of age who are prescribed antibiotics (single or multiple antibiotics, oral or intravenous) will be recruited from the Fargo VAMC Primary Care Clinic area.
* Participants must be able to swallow a capsule.

Exclusion Criteria:

* Exclusion criteria include diarrhea on admission or within the preceding week
* Reported recurrent diarrhea
* Antibiotics in the past four weeks
* Significant underlying conditions (e.g. diabetes, structural cardiac defects including valvular defects, history of infective endocarditis, poor cardiac function, immunosuppression, impaired gut integrity, moderate or serious intestinal disorders, malignancies, pancreatitis, indwelling catheters, recent surgery, recent prolonged hospitalization)
* Previous bowel surgery
* Nutritional restrictions that preclude participation
* Hypersensitivity to penicillin G, ampicillin, or erythromycin
* Persons who have been prescribed their antibiotic for a duration longer than 3 weeks

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea | Approximately one month

CONTACTS AND LOCATIONS:
Locations (1):
- Fargo VA Medical Center, Fargo, North Dakota, United States